CLINICAL TRIAL: NCT05164627
Title: Dexmedetomidine Versus Magnesium Infusion in Reducing Agitations in Pediatric Patients Undergoing Adenotonsillectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, beshoy gamal, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Ain Shams University hospital
Record Dates: First submitted 2021-11-26; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Postoperative Agitations in Pediatric Patients
Keywords: Dexmedetomidine, Magnesium Sulphate, Agitations
MeSH Terms: interventions — Dexmedetomidine; Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): patients will receive Dexmedetomidine infusion (0.2 mcg/kg/hr) from the start of the surgery till the end of it.
  Interventions: Drug: Dexmedetomidine
- Group B (Active Comparator): patients will receive Magnesium infusion (10 mg/kg/hr) from the start of the surgery till the end of it.
  Interventions: Drug: Magnesium Sulphate
- Group C (Placebo Comparator): Patients will receive Normal Saline 0.9% infusion
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — patients will receive Dexmedetomidine infusion (0.2 mcg/kg/hr) from the start of the surgery till the end of it.
  Arms: Group A
Drug: Magnesium Sulphate — patients will receive Magnesium infusion (10 mg/kg/hr) from the start of the surgery till the end of it.
  Other Names: patients will receive Magnesium infusion (10 mg/kg/hr) from the start of the surgery till the end of it.
  Arms: Group B
Drug: Normal saline — After patient arrival at the PACU, Paediatric Anaesthesia Emergence Delirium (PAED) scale ,Ramsay sedation scores (RSS), emergence agitation, HR, and mean arterial blood pressure (MAP) were recorded every 5 min during the first 30 min, then every 10 min for the remaining 30 min of the recovery room stay. Patients were then transferred to the ward. All postoperative observations and scores were performed by the same anesthesiologist who was blinded to the group assignment
  Arms: Group C

SUMMARY:
The aim of this study is evaluating the efficacy and safety of dexmedetomidine versus Magnesium for reducing emergence agitation after adenotonsillectomy in children.

Secondary outcome is to reduce child needs for analgesics and to reduce their dose.

DETAILED DESCRIPTION:
Preoperatively, Intravenous access using EMLA cream will be established in the ward. Child will be introduced to information about GA, OR and surgery. This information will include pictures of the staff and the OR, facemask, blood pressure cuff, etc. The child will move from ward to Pre-Anesthesia Care Unit accompanying his/her parents and anesthesia doctor to establish bonding. Cooperation on induction will be evaluated by using four-point scale with score of 1 to 2 being satisfactory and 3 to 4 being unsatisfactory. If the child develop agitation (Score 3 or 4) emergency Midazolam 0.1 mg/kg IV will be given and the child will be ruled out of study.

Monitors for non-invasive blood pressure, heart rate, electrocardiogram (ECG), pulse oximetry (SpO2) will be attached. Induction of anesthesia will be done using 8% Sevoflurane in oxygen gas with Atracurium 0.5 mg/kg and fentanyl 0.5 mcg/kg to facilitate tracheal intubation. The patients will be divided into three groups:

oGroup A (Dexmedetomidine Group): patients will receive Dexmedetomidine infusion (0.2 mcg/kg/hr) from the start of the surgery till the end of it.

oGroup B (Magnesium Group): patients will receive Magnesium infusion (10 mg/kg/hr) from the start of the surgery till the end of it.

oGroup C (Control Group): Patients will receive Normal Saline 0.9% infusion

Maintenance of anesthesia will be done by using of Sevoflurane 2% in oxygen gas. Controlled mechanical ventilation will be done to maintain normocapnia. Rescue doses of Fentanyl (0.5 mcg/kg) will be given if the patient develop pain. Intraoperative pain is defined as development of Tachycardia (> 20% of baseline heart rate reading) and Hypertension (>20% of Baseline Mean Arterial Blood Pressure reading) .

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II.
* Age group: 4-12 years old.
* The procedure expected to be completed within 1 hour.

Exclusion Criteria:

* Patients with expected difficult airway management.
* lack of consent.
* known adverse effects to dexmedetomidine.
* Mental retardation developmental delay, or neurological or psychiatric illness that may associate with agitation (cerebral palsy, seizure..etc.)
* Hemodynamically unstable patients.
* Persistent cough or high airway secretions.
* Clinical signs of active infectious disease.
* Coagulopathy (INR >1.5).
* Obesity (BMI >30 Kg/m2 ).
* Surgical complication

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-01-08 (Actual); Primary Completion 2022-11-07 (Estimated); Study Completion 2022-12-07 (Estimated)

PRIMARY OUTCOMES:
The Cravero scale. | up to one hour in Post-anesthesia care unit
  it has five steps from obtunded and unresponsive to wild thrashing behaviour requiring restraint. A score of ≥4 (from crying and difficult to console to wild thrashing) for a 5 or more min duration despite active calming efforts is regarded as indicative of ED.
  Behaviour Score Obtunded with no response to stimulation 1 Asleep but responsive to movement or stimulation 2 Awake and responsive 3 Crying (for >3 min) 4 Thrashing behaviour that requires restraint 5
Ramsay sedation scores (RSS) | up to one hour in Post-anesthesia care unit
  1. Patient is anxious and agitated or restless, or both
  2. Patient is co-operative, oriented, and tranquil
  3. Patient responds to commands only
  4. Patient exhibits brisk response to light glabellar tap or loud auditory stimulus
  5. Patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus
  6. Patient exhibits no response

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All IPD sharing plan will be available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: one year

REFERENCES:
- [Result] Shukry M, Clyde MC, Kalarickal PL, Ramadhyani U. Does dexmedetomidine prevent emergence delirium in children after sevoflurane-based general anesthesia? Paediatr Anaesth. 2005 Dec;15(12):1098-104. doi: 10.1111/j.1460-9592.2005.01660.x. PMID 16324031